CLINICAL TRIAL: NCT04793685
Title: Prazosin Treatment for Alcohol Use Disorder With Alcohol Withdrawal Symptoms
Brief Title: Prazosin for Alcohol Use Disorder With Withdrawal Symptoms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000029805; R01AA029113-01 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Withdrawal
MeSH Terms: interventions — Prazosin; Secondary Prevention

STUDY DESIGN:
Intervention Model Description: Patients randomized to Prazosin 16 mg/day titrated over 2 weeks versus placebo taken for 12 weeks with week 12 taper of study medications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Drug (Experimental): Prazosin (16mg/day) versus Placebo comparator, administered in t.i.d schedule, in capsules, over a 12 week period, with 2 weeks titration in weeks 1-2 and a 5-day taper in week 12.
  Interventions: Drug: Prazosin; Behavioral: 12-Step Facilitation with Relapse Prevention and Contingency Management
- Placebo Drug (Placebo Comparator): Placebo for 12 weeks.
  Interventions: Behavioral: 12-Step Facilitation with Relapse Prevention and Contingency Management

INTERVENTIONS:
Drug: Prazosin — Prazosin (16mg/day) versus Placebo comparator, with a 2 week titration period, 9 weeks at full dose and a 5-day taper in week 12.
  Other Names: Minipress
  Arms: Active Drug
Behavioral: 12-Step Facilitation with Relapse Prevention and Contingency Management — 12-Step Facilitation and relapse prevention weekly support and Contingency Management for each weekly appointment to support treatment attendance for all subjects.

SUMMARY:
This is a Phase 2 single site randomized clinical trial (RCT) to be supported by a new NIH-NIAAA grant, R01-AA029113-01, to assess the efficacy of Prazosin (16mg/day) versus Placebo over a 12 week treatment period, followed by a 1- and 3- month assessments post-treatment for individuals with Alcohol Use Disorder (AUD) and history of past or current evidence of alcohol withdrawal symptoms. If medical detoxification is required for any patient, patients would be enrolled after medical detoxification. for those not requiring detoxification, they will be enrolled directly without any requirement of alcohol abstinence. All patients will be provided behavioral counseling weekly with a trained counselor to support recovery during the trial. Primary outcome will be percent of any heavy drinking days and secondary drinking outcomes will be percent of subjects with no heavy drinking days (PSNHDD), avg drinks per drinking day and %of any drinking drinking days as well as additional secondary outcomes of craving, mood and anxiety problems.

DETAILED DESCRIPTION:
In this Phase 2 single site RCT, individuals with moderate to severe alcohol use disorder (AUD) and presence of alcohol withdrawal symptoms (greater than 3 symptoms or more) will be enrolled in a 12 week trial with a 1- and 3- month follow up assessment. Subjects will be randomized to 16 mg /day Prazosin (PR) or Placebo (PBO) with a 2 week titration period and9-week full dose period and week 12 taper. All subjects will be assessed 2X weekly and also provided weekly behavioral counseling to support recovery.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Withdrawal (AW) scores of 3 or more on the CIWA-Ar at treatment entry OR 2 or more Alcohol Withdrawal Syndrome (AWS) symptoms and regular weekly heavy drinking at treatment entry;
* Must meet current DSM-5 criteria for moderate to severe Alcohol Use Disorder (AUD) using SCID-I for DSM-5;
* No health conditions that would impact trial participation as verified by screening and physical examination;
* Able to read English and complete study evaluations
* Able to provide informed written and verbal consent.

Exclusion Criteria:

* Meet current criteria for moderate to severe substance use disorders from use of any another psychoactive substance, excluding nicotine, cocaine and cannabis;
* Current use of illicit /non-prescribed opioids more than 2X/month;
* Regular use of anticonvulsants, sedatives/hypnotics, oral prescription analgesics (other than non-steroidal anti-inflammatory drugs), antiretroviral medications, tricyclic antidepressants, topiramate, baclofen, and regular weekly use of benzodiazepines, as defined by use of three or more times per week;
* Prescribed use of antihypertensive medications that duplicate the mechanism of action at the alpha1 receptor as prazosin or are contraindicated, such as those medications that are also alpha1-adrenergic antagonists (i.e., doxazosin, tamsulosin, terazosin) or are beta-blockers (e.g., propranolol); Potential participants who are prescribed cardiovascular/antihypertensive medications will undergo clinical review by the study PIs and team. Individuals who are prescribed anti-hypertensives that do not duplicate the action of prazosin and are not contraindicated, including ACE inhibitors, angiotensin receptor blockers (ARBs), diuretics, and calcium channel blockers, may be allowed to participate after review from the study physician and principal investigators, with careful monitoring of these individuals' blood pressure at all in-person appointments.
* Psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania);
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study;
* Any psychotic disorder or current Axis I psychiatric disorders requiring specific attention, including need for psychiatric medications;
* Hypotensive individuals with sitting blood pressure below 100/50 mmHG;
* Women who are pregnant, nursing or refuse to use a reliable form of birth control (as assessed by pregnancy tests during initial medical evaluation, and assessed every two weeks during the course of the study).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent Heavy Drinking Days | weeks 3 - 12 of full dose treatment
  Percent of overall days with heavy drinking days (defined by 5 or more drinks per day in men and 4 or more drinks/day in women) after achieving full treatment dose in week 3.

SECONDARY OUTCOMES:
Percent Any Drinking Days | after full dose in weeks 3-12 of treatment period
  Percent of any drinking days over a 12 week period.
Average Drinks per Drinking Day | after full dose in weeks 3-12 treatment period
  The average number of drinks consumed per drinking day assessed weekly over the treatment period.

OTHER OUTCOMES:
Percent of Subjects with no Heavy Drinking Days | weeks 3- 12
  Prazosin versus Placebo treated subjects will be compared on any days of heavy drinking which is defined by 5 or more drinks per day in men and 4 or more drinks/day in women. This will be measured by the Percent of Subjects with no Heavy Drinking Days (PSNHDD) after achieving full dose week 3 through 12 time period.

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, MD, Study Director — Yale University; Gretchen Hermes, MD, Study Director — Yale University
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be uploaded to NIAAA data archive (NIAAA-DA housed within the NIMH Data archive (NDa). as per NIH-NIAAA guidelines.
Supporting Information: SAP, CSR
Time Frame: Baseline data will be uploaded twice yearly. clinical trial outcome data will be shared after study completion and breaking the blind and completion of final analysis of the main study outcomes.
Access Criteria: Access will be provided following the NIH-NIAAA guidelines available at https://grants.nih.gov/grants/guide/notice-files/NOT-AA-19-020.html at the URL below.
URL: http://nda.nih.gov/contribute/contribute-data.html

REFERENCES:
- [Background] Sinha R, Wemm S, Fogelman N, Milivojevic V, Morgan PM, Angarita GA, Hermes G, Fox HC. Moderation of Prazosin's Efficacy by Alcohol Withdrawal Symptoms. Am J Psychiatry. 2021 May 1;178(5):447-458. doi: 10.1176/appi.ajp.2020.20050609. Epub 2020 Nov 19. PMID 33207935